CLINICAL TRIAL: NCT05700643
Title: Effects of Montmorency Cherry Supplementation on Sleep and Inflammatory Outcomes
Brief Title: Montmorency Cherry Supplementation, Sleep, and Inflammation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Cherry Marketing Institute (Unknown)
Responsible Party: Principal Investigator, Robin Tucker, Associate Professor, Michigan State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00008275
Record Dates: First submitted 2022-12-07; First posted 2023-01-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Insomnia Chronic; Inflammation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 500 mg cherry supplement
  Interventions: Dietary Supplement: Montmorency cherry supplement
- Control (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Montmorency cherry supplement — Montmorency cherry supplement
  Arms: Intervention
Dietary Supplement: Control — Placebo
  Arms: Control

SUMMARY:
This study will test the effects of Montmorency cherry supplementation on sleep outcomes and inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) of ≥ 25.0 kg/m2;
* sleep issues as identified by a global score of 5 or greater on the Pittsburgh Sleep Quality Index (PSQI) and/or a score 8 or higher on the Insomnia Severity Index (ISI);
* ability to adhere to a diet low in antioxidants during the study period; and
* willingness to wear a Fitbit for the duration of the study and to wear the Zmachine on selected nights.

Exclusion Criteria:

* unwilling or unable to stop the use of sleep medication
* unable to attend laboratory visits on the East Lansing, Michigan campus

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Change in total sleep time | Through study completion, two weeks for each arm
  sleep duration in hours and minutes
Change in sleep quality | Through study completion, two weeks for each arm
  Pittsburgh Sleep Quality Index scores, scores range from 0-21, higher scores indicate worse outcomes
Change in insomnia symptoms | Through study completion, two weeks for each arm
  Insomnia Severity Index scores, scores range from 0-28, higher scores indicate worse outcomes

SECONDARY OUTCOMES:
Change in C-reactive protein | Through study completion, two weeks for each arm
  blood work
Change in Interleukin-6 | Through study completion, two weeks for each arm
  blood work
Change in Interleukin-8 | Through study completion, two weeks for each arm
  blood work
Change in Interleukin-17 | Through study completion, two weeks for each arm
  blood work
Change in Tumor necrosis factor-alpha | Through study completion, two weeks for each arm
  blood work
Change in Anthropometrics | Through study completion, two weeks for each arm
  Percent body fat

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data available upon request upon completion of analysis.